CLINICAL TRIAL: NCT01439750
Title: Bortezomib (VELCADE), Cladribine and Rituximab (VCR) in Mantle Cell Lymphoma: A Phase I/II Study (PSHCI 10-011)
Brief Title: Bortezomib (VELCADE), Cladribine and Rituximab (VCR) in Mantle Cell Lymphoma (PSHCI 10-011)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Jeffrey J. Pu, MD, PhD, Associate Professor of Medicine, Milton S. Hershey Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSHCI 10-011
Record Dates: First submitted 2011-08-16; First posted 2011-09-23 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Mantle Cell Lymphoma
Keywords: mantle cell lymphoma; lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma | interventions — Rituximab; Bortezomib; Cladribine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Phase I (Experimental): The phase I portion of the study is a standard dose-escalation schemed designed to determine the maximum tolerated dose (MTD) of cladribine in the combination of bortezomib, cladribine, and rituximab therapy. The MTD is defined as the dose level in which ≤1 out of 6 patients have dose-limiting toxicity (DLT). Rituximab 375 mg/m2 on day 5,12, 19, 26 for 1st cycle, then day 5 of cladribine for next 5 cycles and then every 2 months maintenance dose. Cladribine 3-5 mg/m2 days 1-5 for 6 cycles. Bortezomib 1.6 mg/m2 sub Q days 12,19,26 for 3 cycle, then every 2 weeks maintenance dose until toxicity or progression.
  Interventions: Drug: Rituximab; Drug: bortezomib; Drug: Cladribine
- Phase II (Experimental): The phase II portion of the study is a two-arm, single-stage design with no interim analysis. One arm will accrue newly diagnosed patients, and one arm will accrue relapsed patients. In each arm, the progression-free survival rate at 2 years will be used as the primary endpoint for determining whether the treatment is sufficiently active in each arm. No comparisons will be made between the arms. Rituximab 375 mg/m2 on day 5,12,19,26 for 1st cycles, then day 5 montly for next 5 cycles, then every 2 months maintenance dose. Cladribine 3-5 mg/m2 days for 6 cycles (dose determined from phase I). Bortezomib 1.6 mg/m2 weekly on day 12,19,26 for 3 cycles then every 2 weeks as maintenance dose until toxicity or progression.
  Interventions: Drug: Rituximab; Drug: bortezomib; Drug: Cladribine

INTERVENTIONS:
Drug: Rituximab — 375 mg/m2 on day 5, 12, 19, 26 of Cycle1; and day 5 of Cycles 2-6; then every 2 months as maintenenace dose
  Other Names: Rituxam
Drug: bortezomib — 1.6 mg/m2 day 12, 19, 26 for 3 cycles (28 days). Then beginning with Cycle 4, 1.6/mg/m2 every two weeks (Days 5 and 19; maintenance every other week until toxicity or proression of disease).
  Other Names: VELCADE
Drug: Cladribine — Phase I will use 3 dose levels Level 1: caldribine (2-CdA) 3mg/m2 days 1-5; Level 2 caldribine 4mg/m2 days 1-5; Level 3: cladribine 5mg/m2 days 1-5
  Other Names: Litak; Movectro

SUMMARY:
This is a phase I/II trial of bortezomib, cladribine, and rituximab in newly diagnosed and relapsed mantle cell lymphoma (MCL). The phase I component has three dose levels of cladribine (3 mg/m2, 4 mg/m2, and 5 mg/m2) and is designed as a traditional dose-escalation study in which cohorts of 3 patients are evaluated for the incidence of dose-liming toxicity (DLT) at each dose level. Once the maximum tolerated dose (MTD) is determined, a phase II component with 2 arms will begin. One arm will enroll newly diagnosed MCL patients and one arm will enroll relapsed MCL patients. Each arm is a single-stage, fixed sample size study and will be accrued and analyzed separately. The phase I and II data will also be analyzed separately.

DETAILED DESCRIPTION:
The phase I portion of the study is a standard dose-escalation schemed designed to determine the maximum tolerated dose (MTD) of the combination of bortezomib, cladribine, and rituximab therapy. The MTD is defined as the dose level in which ≤1 out of 6 patients have dose-limiting toxicity (DLT). Three patients are enrolled on a dose level. If 0 out of 3 patients have DLT, then the next set of 3 patients are enrolled at the next highest dose level. If ≥2 out of 3 patients have DLT, then the MTD will have been exceeded and dose escalation will cease. Three additional patients will be enrolled at the next lowest dose level if only 3 were treated previously at that level. If 1 out of 3 patients have DLT, then the next set of 3 patients will be treated at the same dose level. If ≤1 out of 6 patients treated at that dose level have DLT, then the next set of patients will be treated at the next higher dose level. If ≥2 out of 6 patients treated at that dose level have DLT, then the MTD will have been exceeded and dose escalation will cease. Three additional patients will be treated at the next lowest dose level if only 3 were treated previously at that level. This phase I study will use 3 dose levels of cladribine (3 mg/m2, 4 mg/m2, and 5 mg/m2), with 3 mg/m2 being the starting dose level. DLTs will be assessed at the completion of the first 2 cycles of cladribine and rituximab.

Phase II Design: The phase II portion of the study is a two-arm, single-stage design with no interim analysis. One arm will accrue newly diagnosed patients, and one arm will accrue relapsed patients. In each arm, the progression-free survival rate at 2 years will be used as the primary endpoint for determining whether the treatment is sufficiently active in each arm. No comparisons will be made between the arms.

Due to difficulties with enrollment, this trial will not move into the intended Phase II of the proposed Phase I/II study. This study will only be Phase I.

ELIGIBILITY:
Inclusion Criteria:

* Females that are postmenopausal for at least 1 year before the screening visit, surgically sterilized or if they are of childbearing potential agree to practice 2 effective methods of contraception from the time of signing the informed consent form through 30 days after the last dose.
* Male subjects must agree to practice effective barrier contraception during the entire study treatment period and through a minimum of 30 days after the last dose of study drug, or completely abstain from heterosexual intercourse.
* Patients with newly diagnosed and relapsed mantle cell lymphoma.
* ECOG performance status grade 3 or higher.

Exclusion Criteria:

* Patient has a platelet count of <50x10 9/L within 14 days before enrollment if not related to disease.
* Patient has an absolute neutrophil count less than 100 within 14 days before enrollment if not related to disease.
* Patient has a calculated or measured creatinine clearance of <20 mL/minute within 14 days before enrollment.
* Patient has > Grade 2 peripheral neuropathy within 14 days before enrollment.
* Patient has > 1.5 x ULN total bilirubin.
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association Class II or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Patient has hypersensitivity to bortezomib, boron or mannitol.
* Female subject is pregnant or breast-feeding.
* Patient has received other investigational drugs within 14 days before enrollment.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Dose Limiting Tolerability | 2 years
  Dose Limiting Tolerability as measured by CTCAEv.4 criteria and to evaluate progression free survival in patients treated with VCR in the Phase 1 portion .

SECONDARY OUTCOMES:
Secondary Outcome objective response rates | 7 months
  Estimate objective response rates of the VCR regimen in B cell malignancies where response to therapy is assessed per the revised Cheson criteria (2007) and the overall survival of patients treated with this combination for the Phase 2 portion of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J Pu, MD PhD, Principal Investigator — Milton S. Hershey Medical Center
Locations (2):
- United States (2):
  - Penn State Cancer Institute, Hershey, Pennsylvania
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided
May share data

REFERENCES:
- [Derived] Pu JJ, Berger KN, Zheng C, Do N, Claxton DF, Ehmann WC, Drabick JJ, Li H, Loughran TP Jr, Epner EM. A phase I study using bortezomib (Velcade), cladribine, and rituximab in treating patients over 50 years old with mantle cell lymphoma. Front Oncol. 2024 Dec 16;14:1449401. doi: 10.3389/fonc.2024.1449401. eCollection 2024. PMID 39737396